CLINICAL TRIAL: NCT01566656
Title: Allogeneic Hematopoietic Stem Cell Transplantation Using a Non-myeloablative Preparative Regimen of Total Lymphoid Irradiation and Anti-thymocyte Globulin for Older Patients With Relapsed Lymphoid Malignancies
Acronym: TLI-ATG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRD/10/06-L
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Haemato-lymphoid Malignancies or Syndromes in Whom Allogeneic Stem Cell Transplantation is Warranted
Keywords: Allogeneic hematopoietic stem cell transplantation; Non-myeloablative preparative regimen; Total lymphoid irradiation; Anti-thymocyte globulin; Lymphoid malignancies
MeSH Terms: interventions — Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TLI and anti-thymocyte globulin (Experimental)
  Interventions: Drug: total lymphoid irradiation and anti-thymocyte globulin

INTERVENTIONS:
Drug: total lymphoid irradiation and anti-thymocyte globulin — * TLI Administration: TLI is administered ten times in 120 cGy fractions on day -11 through day -7 and day -4 through day -1.
  * ATG: Thymoglobulin will be administered five times intravenously at 1.5 mg/kg/day from day -11 through day -7 for a total dose of 7.5 mg/kg.
  * Mobilized PBSCs (Day 0): The desired cell doses (based on recipient body weight) for MRD and MUD transplants are around 4-8 x106 CD34+ cells/kg.
  * GVHD Prophylaxis: Cyclosporine A (CSP) 3 mg/kg IV from day-3 and Mycophenylate mofetil (MMF) 500 mg x 4/ day PO from day 0

SUMMARY:
Recent advances in allogeneic hematopoietic cell transplantation (allo-SCT) have led to reduce intensity preparative regimens that are non-myeloablative and reduce the toxicities associated with the transplant. Consequently non-relapse mortality has been reduced, including in elderly patients with comorbidities. However, despite this benefit in terms of toxicity, excessive reduction of the intensity preparative regimens may favor relapse of the initial illness. Thus, acute and chronic graft-versus-host disease and opportunistic fungal and viral infections are always serious complications. The aim of our study is to check if a new modality of reduced intensity preparative regimen combining total lymphoid irradiation (TLI) and thymoglobulin (ATG), would limit the toxicity of treatment and reduce the incidence of acute GVHD after allogeneic transplantation while preserving the antitumor benefit.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with one of the following hemato-lymphoid malignancies or syndromes in whom allogeneic stem cell transplantation is warranted. Specific disease categories include: non-follicular indolent advanced stage Non-Hodgkin Lymphomas, Mantle Cell Lymphoma, Marginal zone lymphoma, MALT, T cell lymphoma, Chronic Lymphocytic or prolymphocytic Leukemia, Hodgkin Disease, and Waldenström macroglobulinemia. T-cell NOS, angioimmunoblastic lymphoma, HTLV1, T-gamma/delta, anaplastic lymphoma and Sezeay syndromes can be included after careful assessment by the PI and the protocol steering committee.
* Patients must be at least in partial remission (according to standard criteria) after salvage therapy and before (~one month) the start of the conditioning regimen.
* Patient age >50 and less than 66 years, or for patients <50 years of age but because of pre-existing medical conditions or prior therapy are considered to be at high risk for regimen-related toxicity associated with conventional myeloablative transplants.
* A fully HLA-identical sibling or matched unrelated donor is available (10/10 HLA match). Patients with one antigen mismatched donors can be considered but only after discussion with the transplant team and the Principal Investigator.
* Patient must be competent to give consent.

Exclusion Criteria:

* Patients with progressive hematolymphoid malignancies despite conventional therapies, and not in partial remission during the month preceding transplantation.
* Patients with DLBCL or cutaneous T cell lymphoma
* Uncontrolled CNS involvement with disease
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Females who are pregnant
* Organ dysfunction defined as follows:
* Cardiac function: ejection fraction <30% or uncontrolled cardiac failure
* Pulmonary: DLCO <40% predicted
* Renal: Serum creatinine >1.0 mg/dL; if serum creatinine >1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be >60 mL/min/1.73 m²
* Liver function abnormalities: elevation of bilirubin to > 3 mg/dl and/or transaminases >4x the upper limit of normal
* Karnofsky performance score < 70%
* Patients with poorly controlled hypertension on multiple antihypertensives
* Documented fungal disease that is progressive despite treatment
* Viral infections: HIV positive patients. Hepatitis B and C positive patients will be evaluated on a case by case basis
* Psychiatric disorders or psychosocial problems which in the opinion of the primary physician or Principal Investigator would place the patient at unacceptable risk from this regimen.
* Patients with prior malignancies diagnosed > 5 years ago without evidence of disease are eligible. Patients with a prior malignancy treated < 5 years ago but have a life expectancy of > 5 years for that malignancy are eligible.

Ages: 50 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-03-02 (Actual); Primary Completion 2016-11-29 (Actual); Study Completion 2016-11-29 (Actual)

PRIMARY OUTCOMES:
To evaluate the incidence of non-relapse mortality (NRM) | one year after transplantation

SECONDARY OUTCOMES:
Neutrophil and platelets recovery and chimerism measurement
  To evaluate the kinetics of donor hematopoietic cell engraftment (neutrophil and platelets recovery) and chimerism.
T cell subsets, regulatory cells, NK cells and B cells measurement
  To document the quantitative and qualitative reconstitution of the immune system including T cell subsets, regulatory cells, NK cells and B cells.
Number of relapse, acute and chronic GVHD | one year after transplantation
  To evaluate the rate of relapse, overall and event-free survival and incidence of acute and chronic GVHD, at one year after transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad MOHTY, Pr, Principal Investigator — Hôpital Saint Antoine (AP-HP)
Locations (4):
- France (4):
  - Besançon University Hospital, Besançon
  - Lille University Hospital, Lille
  - Lyon University Hospital, Lyon
  - Nantes University Hospital, Nantes